CLINICAL TRIAL: NCT03581396
Title: Scleral Hydrops and Intralabyrinthine Schwannoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7026
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Hydrops Saccular
Keywords: Hydrops sacculaire; schwannoma intralabyrinth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The symptoms of intralabyrinthine schwannomas (vertigo, deafness, instability, tinnitus) cut across the symptoms found in pressure pathologies involving the inner ear, particularly the endolymphatic hydrops.

Some publications have described dilatation of the membranous labyrinth (hydrops) in the presence of intralabyrinthine tumors.

It would be interesting to measure the size of the saccule (structure of the membranous labyrinth) in the presence of an intralabyrinthine schwannoma, to evaluate if some of the symptoms presented by the patients could be explained by the concomitant presence of an endolymphatic hydrops (accessible to drug therapy - Betahistine).

ELIGIBILITY:
Inclusion Criteria

* Age> 18,
* Subject having benefited from an exploration of internal auditory canals by MRI in our service at CHU de Hautepierre between January 1, 2008 and October 1, 2017
* Presence on the MRI of the internal auditory ducts, including the realization of a high resolution fluid sequence of FIESTA-C (exploitable) type, of an intralabyrinthine schwannoma, without extension to the internal auditory canal.
* Subject who has agreed to the use of medical data for the purposes of this research.

Criteria for Non Inclusion

* Refusal of the patient to participate in the study
* Absence of high resolution fluid sequence of fast imaging employing steady state acquisition (FIESTA-C)
* Presence of movement artifacts interfering with the interpretation of the FIESTA-C sequence
* Interior surgery of the inner ear or pontocerebellar angle, without preoperative imaging Inflammatory or infectious pathology of the concomitant middle or inner ear
* Extension of schwannoma to the internal auditory canal
* Impossibility of giving the subject informed information (difficulty understanding the subject,)
* Subject under the protection of justice
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having benefited from an exploration of internal auditory canals by MRI in our service at CHU de Hautepierre between January 1, 2008 and October 1, 2017
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Size of intralabyrinth saccules | 1 hour after the realization of the MRI]
  To measure saccule size (membranous labyrinth structure) in patients with intralabyrinthine schwannoma on a high resolution fluid sequence (FIESTA-C) in 3T MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Service Imagerie 1, Strasbourg, France